CLINICAL TRIAL: NCT03751280
Title: A Randomized, Sham-Controlled Study of PEAR-004 as an Adjunct to Standard-of-care Treatment for Schizophrenia
Brief Title: Study of Efficacy of PEAR-004 in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPEA001A12201
Record Dates: First submitted 2018-11-08; First posted 2018-11-23 (Actual); Results first posted 2020-11-23 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Digital Therapeutic; CBT; smartphone app; mental disorder; psychosis; acute psychotic reaction; chronic psychosis; failure to recognize what is real; false beliefs; unclear thinking,; confused thinking; auditory hallucinations; paranoia; reduced social engagement; reduced emotional expression
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Psychotic Disorders; Hallucinations; Paranoid Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- PEAR-004 (Experimental): Eligible participants were able to access PEAR-004 (an investigational digital therapeutic) on a mobile device (iOS and Android based) as needed to receive suggestions about coping strategies to overcome difficulties in daily life.
  Interventions: Device: PEAR-004
- Sham (Sham Comparator): Eligible participants were able to access a sham control downloaded on a mobile device (iOS and Android based) as needed to receive notifications prompting the participant to open the sham app, which displayed a prescription timer for the remaining duration of app availability.
  Interventions: Device: Sham

INTERVENTIONS:
Device: PEAR-004 — PEAR-004 (an investigational digital therapeutic) or sham (control) was downloaded to the subject's phone and then the assigned application was unlocked using a prescription code provided by Pear Therapeutics. As this was a digital therapeutic device study, dose or mode of administration is not applicable.
  Arms: PEAR-004
Device: Sham — PEAR-004 (an investigational digital therapeutic) or sham (control) was downloaded to the subject's phone and then the assigned application was unlocked using a prescription code provided by Pear Therapeutics. As this was a digital therapeutic device study, dose or mode of administration is not applicable.
  Arms: Sham

SUMMARY:
The purpose of the study was to determine in patients currently being administered antipsychotic pharmacotherapy whether PEAR-004 could further reduce symptoms of schizophrenia as measured by the Positive and Negative Syndrome Scale (PANSS).

The overall rationale for the study was to assess the first prescription digital therapeutic (PDT) in schizophrenia using a form of proven psychosocial intervention, cognitive behavioral therapy (CBT), to supplement standard of care with antipsychotic medications.

DETAILED DESCRIPTION:
This was a randomized, sham-controlled, rater-blinded, parallel group trial. Overall, 112 subjects were randomized 1:1 in to the following groups:

* Group A: Clinician-directed pharmacotherapy + PEAR-004
* Group B: Clinician-directed pharmacotherapy + sham app An up to 28-day screening period included standard screening assessments as defined in the assessment schedule. Eligible subjects were randomized on Day 1 into one of the treatment groups.

Subjects in both groups continued to receive their clinician-directed standard-of-care treatment for schizophrenia, including pharmacotherapy. Subjects in Group A used PEAR 004 and subjects in Group B used a sham for a period of 12 weeks. Subjects returned to the clinic for outpatient visits at Week 4 (day 29), Week 8 (day 57), and Week 12 (day 85). At each visit, standard assessments were performed according to the assessment schedule, including PANSS, ISST-Plus, CGI, BMQ, MAP-SR, WHOQOL-BREF, BDI-II, ISI, and adverse events (AEs). A final follow-up visit was performed at Week 16 (day 115),

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Healthy male and female subjects 18 to 65 years of age, inclusive, and in good health as determined by medical history, physical examination, and vital signs at screening
* SCID-based DSM-5 diagnosis of schizophrenia and a total PANSS score > 60
* Proficient in English at 5th grade reading level or higher, in the judgement of the investigator
* Capable of using a mobile device (compatible with PEAR-004) and using common applications, in the judgement of the investigator

Key Exclusion Criteria:

* Major change in primary antipsychotic medication in the prior 4 weeks before screening (e.g., switching to a new agent or a dose adjustment within two weeks of randomization)
* Planning to move out of the geographic area within 3 months
* Unable to use English to participate in the consent process, the interventions or assessments
* Inability to comply with study procedures, due to severe medical conditions or otherwise
* Meet DSM-5 diagnosis for a current episode of major depression, mania, or hypomania in the past month
* Meet DSM-5 diagnosis for a current moderate or severe alcohol or cannabis use disorder in the past 2 months
* Meet DSM-5 diagnosis for a current substance use disorder (other than alcohol or cannabis) in the past 2 months
* Considered high risk for suicidal behavior based on ISST-Plus score at screening, or in the judgement of the investigator
* Previously participated in a clinical study involving PEAR-004

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (6):
  - Novartis Investigative Site, Garden Grove, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Maitland, Florida
  - Novartis Investigative Site, Grand Rapids, Michigan
  - Novartis Investigative Site, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Ghaemi SN, Sverdlov O, van Dam J, Campellone T, Gerwien R. A Smartphone-Based Intervention as an Adjunct to Standard-of-Care Treatment for Schizophrenia: Randomized Controlled Trial. JMIR Form Res. 2022 Mar 28;6(3):e29154. doi: 10.2196/29154. PMID 35343910
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 6 centers in the USA.
Pre-assignment Details: The eligible subjects were randomized in 1:1 ratio to receive either PEAR-004 or sham.
Groups:
- PEAR-004: Eligible participants were to access PEAR-004 (an investigational digital therapeutic) on a mobile device (iOS and Android based) as needed to receive suggestions about coping strategies to overcome difficulties in daily life.
- Sham: Eligible participants were to access a sham control downloaded on a mobile device (iOS and Android based) as needed to delivering notifications prompting the participant to open the sham app, and then display a prescription timer for the remaining duration of app availability.
Period: Overall Study
Arm/Group | PEAR-004 | Sham
Started (All enrolled participants were in Randomized Set) | 56 | 56
Full Analysis Set (FAS) | 54 | 55
Safety Set (SAF) | 55 | 55
Completed | 48 | 44
Not Completed | 8 | 12
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 3 | 5
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set = all randomized participants who received the study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | PEAR-004 | Sham | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (10.99) | 45.7 (11.60) | 44.7 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 36 | 36 | 72
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 3 | 4 | 7
  Black or African American | 28 | 25 | 53
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White | 18 | 25 | 43
  Other | 3 | 0 | 3
Disease duration at baseline [Mean (Standard Deviation); unit: Years] — Disease Duration at baseline: Duration (in Years) from informed consent to date of diagnosis. Date of diagnosis corresponds to date where subjects reported schizophrenia diagnosis in medical history at screening visit.
  Years | 16.2 (11.40) | 18.2 (11.56) | 17.2 (11.47)
Total Positive and Negative Syndrome Scale (PANSS) score at baseline [Mean (Standard Deviation); unit: Score] — The Positive and Negative Syndrome Scale (PANSS) assesses: positive (hallucinations, delusions, thought disorder), negative (blunted affect, abstract thinking and general symptomatology. The positive and negative subscale each consist of 7 items rated from 1(absent) - 7(extreme) with a minimum score = 7, maximum score = 49. The general subscale consists of 16 items with a minimum score = 16, maximum score = 112. A Total PANSS score (positive+ negative + general scores) has a minimum of 30 and maximum of 210. Higher scores represent more severity in symptoms.
  Score | 73.5 (10.25) | 72.7 (10.10) | 73.1 (10.14)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Positive and Negative Syndrome Scale (PANSS) Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a well validated, standardized method of evaluating and monitoring psychotic symptoms. The PANSS assesses: positive (hallucinations, delusions, thought disorder), negative (blunted affect, abstract thinking and general symptomatology. The positive and negative subscale each consist of 7 items rated from 1(absent) - 7(extreme) with a minimum score = 7, maximum score = 49. The general subscale consists of 16 items with a minimum score = 16, maximum score = 112. A Total PANSS score (positive+ negative + general scores) has a minimum of 30 and maximum of 210. Higher scores represent more severity in symptoms.
Time Frame: Baseline, Day 29, Day 57, Day 85
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 54 | 55
Score
  Day 29: number analyzed (Participants) | 52 | 54
  Day 29 | -1.6 (0.86) | -2.2 (0.84)
  Day 57: number analyzed (Participants) | 49 | 47
  Day 57 | -2.5 (0.9) | -3.3 (0.9)
  Day 85: number analyzed (Participants) | 48 | 49
  Day 85 | -2.6 (1.14) | -5.3 (1.13)
Statistical Analysis 1: Comparison: PEAR-004 vs Sham; Day 29; Test type: Other; Comparison of adjusted least square mean = 0.61, 90% CI 2-sided [-1.4 to 2.6], Standard Error of Mean 1.200 — mixed effects model with treatment, visit as fixed effects, baseline and disease duration at baseline as continuous covariates, treatment * visit and baseline * visit interaction effects
Statistical Analysis 2: Comparison: PEAR-004 vs Sham; Day 57; Test type: Other; Comparison of adjusted least square mean = 0.80, 90% CI 2-sided [-1.3 to 2.9], Standard Error of Mean 1.279 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEAR-004 vs Sham; Day 85; Test type: Other; p = 0.0931, t-test, 2 sided; Comparison of adjusted least square mean = 2.73, 90% CI 2-sided [0.1 to 5.4], Standard Error of Mean 1.611 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Percent of Dropout
Description: Dropout rate to evaluate retention to assigned study treatment
Time Frame: Day 115
Population: Randomized Set
Measure: Count of Participants; unit: Participants
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 56 | 56
Participants | 8 | 12

3. Secondary Outcome: Change From Baseline in the Positive PANSS Score
Description: The PANSS includes 3 scales and 30 items: 7 items that make up the Positive Scale (eg, delusions, conceptual disorganization, hallucinatory behavior); 7 items that make up the Negative Scale (eg, blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal); and 16 items that make up the General Psychopathology Scale (eg, somatic concern, anxiety, guilt feelings, mannerisms and posturing, motor retardation, uncooperativeness, disorientation, poor impulse control, preoccupation). Individual items are scored with values ranging from 1 to 7. Total Negative and Positive Subscale scores each range from 7 to 49; higher score indicates greater severity.
Time Frame: Baseline, Day 29, Day 57, Day 85
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 54 | 55
Score
  Day 29: number analyzed (Participants) | 52 | 54
  Day 29 | -0.2 (0.36) | -0.4 (0.35)
  Day 57: number analyzed (Participants) | 49 | 47
  Day 57 | -0.8 (0.38) | -1.4 (0.38)
  Day 85: number analyzed (Participants) | 48 | 49
  Day 85 | -1.0 (0.46) | -1.8 (0.45)
Statistical Analysis 1: Comparison: PEAR-004 vs Sham; Day 29; Test type: Other; Comparison of adjusted least square mean = 0.21, 90% CI 2-sided [-0.6 to 1], Standard Error of Mean 0.501 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PEAR-004 vs Sham; Day 57; Test type: Other; Comparison of adjusted least square mean = 0.61, 90% CI 2-sided [-0.3 to 1.5], Standard Error of Mean 0.538 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEAR-004 vs Sham; Day 85; Test type: Other; p = 0.2069, t-test, 2 sided; Comparison of adjusted least square mean = 0.82, 90% CI 2-sided [-0.3 to 1.9], Standard Error of Mean 0.648 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in the General Psychopathology PANSS Score
Description: The PANSS includes 3 scales and 30 items: 7 items that make up the Positive Scale (eg, delusions, conceptual disorganization, hallucinatory behavior); 7 items that make up the Negative Scale (eg, blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal); and 16 items that make up the General Psychopathology Scale (eg, somatic concern, anxiety, guilt feelings, mannerisms and posturing, motor retardation, uncooperativeness, disorientation, poor impulse control, preoccupation). Individual items are scored with values ranging from 1 to 7. Total General Psychopathology Subscale score range from 16 to 112; higher score indicates greater severity.
Time Frame: Baseline, Day 29, Day 57, Day 85
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 54 | 55
Score
  Day 29: number analyzed (Participants) | 52 | 54
  Day 29 | -0.8 (0.61) | -1.4 (0.59)
  Day 57: number analyzed (Participants) | 49 | 47
  Day 57 | -1.4 (0.63) | -1.5 (0.63)
  Day 85: number analyzed (Participants) | 48 | 49
  Day 85 | -1.2 (0.76) | -2.8 (0.75)
Statistical Analysis 1: Comparison: PEAR-004 vs Sham; Day 29; Test type: Other; Comparison of adjusted least square mean = 0.51, 90% CI 2-sided [-0.9 to 1.9], Standard Error of Mean 0.849 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PEAR-004 vs Sham; Day 57; Test type: Other; Comparison of adjusted least square mean = 0.12, 90% CI 2-sided [-1.4 to 1.6], Standard Error of Mean 0.890 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEAR-004 vs Sham; Day 85; Test type: Other; p = 0.1368, t-test, 2 sided; Comparison of adjusted least square mean = 1.61, 90% CI 2-sided [-0.2 to 3.4], Standard Error of Mean 1.071

5. Secondary Outcome: Change From Baseline in the Negative PANSS Score
Description: as for outcome 3
Time Frame: Baseline, Day 29, Day 57, Day 85
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 54 | 55
Score
  Day 29: number analyzed (Participants) | 52 | 54
  Day 29 | -0.5 (0.31) | -0.4 (0.3)
  Day 57: number analyzed (Participants) | 49 | 47
  Day 57 | -0.3 (0.32) | -0.5 (0.32)
  Day 85: number analyzed (Participants) | 48 | 49
  Day 85 | -0.4 (0.41) | -0.9 (0.41)
Statistical Analysis 1: Comparison: PEAR-004 vs Sham; Day 29; Test type: Other; Comparison of adjusted least square mean = -0.13, 90% CI 2-sided [-0.8 to 0.6], Standard Error of Mean 0.430 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PEAR-004 vs Sham; Day 57; Test type: Other; Comparison of adjusted least square mean = 0.15, 90% CI 2-sided [-0.6 to 0.9], Standard Error of Mean 0.453 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEAR-004 vs Sham; Test type: Other; p = 0.3798, t-test, 2 sided; Comparison of adjusted least square mean = 0.51, 90% CI 2-sided [-0.5 to 1.5], Standard Error of Mean 0.581 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in the Motivation and Pleasure Self-report (MAP-SR) Score
Description: The MAP-SR is a 15-item self-report measure that provides a total score index of current motivation/pleasure negative symptoms. Responses are given on a 5-point scale where 0 = no pleasure or motivation and 4 = extreme pleasure or motivation. Total scores range from 0 to 60 and higher scores indicate greater motivation and pleasure during everyday activities.
Time Frame: Baseline, Day 29, Day 57, Day 85
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 54 | 55
Score
  Day 29: number analyzed (Participants) | 51 | 54
  Day 29 | 0.8 (1.05) | 1.6 (1.02)
  Day 57: number analyzed (Participants) | 49 | 47
  Day 57 | -0.5 (1.41) | 1.1 (1.43)
  Day 851.43: number analyzed (Participants) | 48 | 49
  Day 851.43 | -1.2 (1.26) | 2.8 (1.25)
Statistical Analysis 1: Comparison: PEAR-004 vs Sham; Day 29; Test type: Other; Comparison of adjusted least square mean = -0.79, 90% CI 2-sided [-3.2 to 1.6], Standard Error of Mean -0.79 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PEAR-004 vs Sham; Day 57; Test type: Other; Comparison of adjusted least square mean = -1.60, 90% CI 2-sided [-4.9 to 1.7], Standard Error of Mean 2.006 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEAR-004 vs Sham; Day 85; Test type: Other; p = 0.0245, t-test, 2 sided; Comparison of adjusted least square mean = -4.07, 90% CI 2-sided [-7.0 to -1.1], Standard Error of Mean 1.780 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in the World Health Organization Quality of Life (WHOQOL-BREF) Scale
Description: The WHOQOL-BREF is a 26-item, self-report questionnaire and short version of WHOQOL-100, consisting of 4 domains: physical health (7 items) (Domain 1), psychological health (6 items) (Domian 2), social relationships (3 items) (Domain 3), and environmental health (8 items) (Domain 4); it also contains QOL and general health items. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). The mean score of items within each domain is used to calculate the domain score. Each individual item of the WHOQOL-BREF is scored from 1=not at all to 5=completely on a response scale, which is stipulated as a 5-point ordinal scale. The scores are then transformed linearly to a scale of 0 (the worse quality of life) to 100 (the worse quality of life).
Time Frame: Baseline, Day 29, Day 57, Day 85
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 54 | 55
Score
  Day 29-Domain 1: number analyzed (Participants) | 52 | 54
  Day 29-Domain 1 | -0.1 (0.37) | 0.1 (0.36)
  Day 57-Domain 1: number analyzed (Participants) | 49 | 47
  Day 57-Domain 1 | -0.3 (0.44) | -0.3 (0.45)
  Day 85-Domain 1: number analyzed (Participants) | 48 | 49
  Day 85-Domain 1 | 0.2 (0.45) | 0.1 (0.45)
  Day 29-Domain 2: number analyzed (Participants) | 52 | 54
  Day 29-Domain 2 | -0.6 (0.4) | -0.1 (0.39)
  Day 57-Domain 2: number analyzed (Participants) | 49 | 47
  Day 57-Domain 2 | -0.7 (0.37) | -0.6 (0.38)
  Day 85-Domain 2: number analyzed (Participants) | 48 | 49
  Day 85-Domain 2 | -0.5 (0.43) | 0.1 (0.42)
  Day 29-Domain 3: number analyzed (Participants) | 52 | 54
  Day 29-Domain 3 | -0.3 (0.28) | 0.1 (0.27)
  Day 57-Domain 3: number analyzed (Participants) | 49 | 47
  Day 57-Domain 3 | -0.3 (0.33) | 0.1 (0.33)
  Day 85-Domain 3 | 0.5 (0.33) | 0.3 (0.33)
  Day 29-Domain 4: number analyzed (Participants) | 52 | 54
  Day 29-Domain 4 | -0.2 (0.61) | -0.9 (0.6)
  Day 57-Domain 4: number analyzed (Participants) | 49 | 47
  Day 57-Domain 4 | -0.5 (0.61) | -0.7 (0.61)
  Day 85-Domain 4 | -0.1 (0.69) | 1.1 (0.68)
Statistical Analysis 1: Comparison: PEAR-004 vs Sham; Day 29-Domain 1; Test type: Other; Comparison of adjusted least square mean = -0.18, 90% CI 2-sided [-1.0 to 0.7], Standard Error of Mean 0.516 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in the Beck Depression Inventory, Second Ed. (BDI-II) Total Score
Description: Beck Depression Inventory (BDI) is a 21-items self reported inventory with a scale evaluating depressive symptoms and the changes in BDI after treatment compared to baseline. The range of scores is 0 to 63, with higher scores indicating greater severity of depression.
Time Frame: Baseline, Day 29, Day 57, Day 85
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 54 | 55
Score
  Day 29: number analyzed (Participants) | 52 | 54
  Day 29 | -1.0 (1.13) | -0.1 (1.11)
  Day 57: number analyzed (Participants) | 49 | 47
  Day 57 | -4.8 (1.14) | -1.5 (1.15)
  Day 85: number analyzed (Participants) | 48 | 49
  Day 85 | -3.4 (1.32) | -3.2 (1.3)

9. Secondary Outcome: Percentage Change From Baseline in Total PANSS Score (Within Assigned Treatment Group)
Description: as for outcome 1
Time Frame: Baseline, Day 29, Day 57, Day 85
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 54 | 55
Score
  Day 29: number analyzed (Participants) | 52 | 54
  Day 29 | -2.0 (1.21) | -3.0 (1.18)
  Day 57: number analyzed (Participants) | 49 | 47
  Day 57 | -3.6 (1.28) | -4.4 (1.29)
  Day 85: number analyzed (Participants) | 48 | 49
  Day 85 | -3.7 (1.57) | -7.1 (1.55)

10. Secondary Outcome: Percentage of Responders as Assessed by the Brief Medication Questionnaire (BMQ)
Description: The Brief Medication Questionnaire (BMQ) collects information about current schizophrenia medication use.
Time Frame: Day 29, Day 57, and Day 85
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 54 | 55
Participants
  Day 1 | 53 | 54
  Day 29 | 52 | 53
  Day 57 | 49 | 46
  Day 85 | 48 | 48
  Day 115 / End of Study | 54 | 52

11. Secondary Outcome: Percentage of Responders as Assessed by the Total PANSS Score
Description: A Response is defined as a reduction of at least 20% at day 85 or last visit in total PANSS score relative to Baseline.
Time Frame: Day 85
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 54 | 55
Participants | 2 | 9

12. Secondary Outcome: Number of Patients With Adverse Events
Description: Adverse events, serious adverse events, and adverse events leading to discontinuation throughout the study
Time Frame: Day 115
Population: Safety Set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 55 | 55
Participants
  Participants with at least one AE | 12 | 10
  Study drug-related AEs | 1 | 0
  Participants with at least one SAE | 0 | 1
  AEs leading to discontinuation of study treatment | 0 | 0
  Study-drug related AEs leading to treatment disc. | 0 | 0

13. Secondary Outcome: Number of Patients With Vital Sign Measurements
Description: Vital signs at baseline, day 85 or last visit
Time Frame: Day 85
Measure: Number; unit: Number of participants
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 55 | 55
Number of participants | 55 | 55

14. Secondary Outcome: InterSePT Scale for Suicidal Thinking-Plus (ISST-Plus) Score
Description: InterSePT Scale for Suicidal Thinking-Plus (ISST-Plus) score. Semi-structured interview to assess severity of suicidal ideation and behavior Part I: collects information on 7 days prior to visit; 13 items scored 0 (min) to 2 (max) for suicidality, with a higher score representing a worse outcome Part II: collects information on suicidal behavior since last visit, with nominal categories Yes / No / Unknown (NA) Part III: global rating of status at time of interview; scored 0 (min) to 5 (max) for suicidality, with a higher score representing a worse outcome.
  Please note that only part III score (severity of suicidal risk) was summarized and reported.
Time Frame: Baseline, Day 29, 57, 85, and 115
Population: The number of subjects analyzed at different visits may differ from the overall number analyzed within a treatment group because some patients missed some visits.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PEAR-004 | Sham
Number analyzed (Participants) | 54 | 53
scores on a scale
  Baseline: number analyzed (Participants) | 52 | 50
  Baseline | 0.0 (0.00) | 0.1 (0.24)
  Day 1: number analyzed (Participants) | 50 | 52
  Day 1 | 0.1 (0.31) | 0.0 (0.14)
  Day 29: number analyzed (Participants) | 51 | 53
  Day 29 | 0.0 (0.28) | 0.1 (0.41)
  Day 57: number analyzed (Participants) | 47 | 46
  Day 57 | 0.1 (0.44) | 0.0 (0.00)
  Day 85: number analyzed (Participants) | 48 | 49
  Day 85 | 0.1 (0.45) | 0.1 (0.32)
  Day 115 / End Of Study | 0.1 (0.43) | 0.1 (0.45)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 119 days.
Groups:
- Total: Total
Arm/Group | PEAR-004 | Sham | Total
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/55 | 1/55 | 1/110
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEAR-004 (N=55) | Sham (N=55) | Total (N=110)
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT03751280/SAP_000.pdf
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT03751280/Prot_001.pdf